CLINICAL TRIAL: NCT00751296
Title: A Phase 2 Study of Lenalidomide in Previously Untreated, Symptomatic Chronic Lymphocytic Leukemia (CLL)
Brief Title: Study of Lenalidomide in Previously Untreated, Symptomatic Chronic Lymphocytic Leukemia (CLL)
Acronym: Rev-CLL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Seven years of follow-up & final analysis done in Dec 2012.
Sponsor: University Health Network, Toronto (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rev-06-0099; RV-CLL-PI-0099 (Other: Study sponsor)
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Results first posted 2016-05-12 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Lymphocytic Leukaemia
Keywords: Lenalidomide; immunomodulatory drug (IMiD®); Thalidomide analogues
MeSH Terms: conditions — Leukemia, B-Cell | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidiomide (Experimental): Lenalidomide target dose of 10 mg PO OD X 3 weeks (days 1-21) followed by 1 week off therapy (days 22-28) on a 28-day cycle.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Subjects will receive lenalidomide, starting at 2.5 mg daily x 3 weeks (days 1-21) and escalating up to a target dose of 10 mg daily X 3 weeks (days 1-21) followed by 1 week off therapy (days 22-28) on a 28 day cycle.Patients will be treated with lenalidomide until disease progression or 2 cycles past CR. (no maximum of cycles).
  Other Names: REVLIMID®

SUMMARY:
This study will assess the

* efficacy (response rate) of oral lenalidomide in the treatment of patients with symptomatic, previously untreated, chronic lymphocytic leukemia (CLL),
* toxicity of lenalidomide in patients with CLL as well as time to progression, stable disease duration and, if responses are observed, response duration.

DETAILED DESCRIPTION:
This is a phase II, nonrandomized, single institution study in symptomatic, previously untreated CLL patients. Subjects will receive the study drug, lenalidomide, starting at 2.5 mg daily x 3 weeks (days 1-21) and escalating up to a target dose of 10 mg daily X 3 weeks (days 1-21) followed by 1 week off therapy (days 22-28) on a 28 day cycle. Although a maximal dose of 10 mg daily (days 1-21) will be targeted, if a patient is felt by the investigator to be benefiting from doses less than the target dose (i.e. 2.5 mg or 5 mg daily), the investigator may at his discretion choose to hold the patient at that dose without further escalation. For those patients who have progressive disease after cycle 3, further dose escalations as assessed by response and toxicity at the end of each escalated dose cycle to a maximum of 25 mg (days 1-21) will be allowed. Patients will be treated with lenalidomide until disease progression or 2 cycles past CR. (no maximum of cycles).

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Age ≥18 years at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* A confirmed diagnosis of B-cell CLL by NCI Working Group criteria
* No prior systemic therapy for CLL. Steroid therapy alone for autoimmune cytopenias (anemia or thrombocytopenia) is NOT considered a prior systemic therapy.
* Radiation: Patients may have received prior radiation therapy restricted to ≤ 25% of functioning bone marrow. Patients must be ≥ 4 weeks since last treatment with radiation therapy.
* Surgery: previous surgery is permissible. Patient must be ≥ 4 weeks since any major surgery.
* Patients must have symptomatic disease requiring therapy. One or more of the following must be present to be eligible:

  * Symptomatic lymphadenopathy
  * Hepatomegaly and/or splenomegaly
  * Anemia (Hb <110 g/L)
  * Thrombocytopenia (platelets <100)
  * Fatigue, weight loss, night sweats, fever (without infection) or other constitutional symptoms felt to require treatment as per treating physician discretion
  * Persistent rise in lymphocyte count with doubling time of < 12 months
* ECOG performance status of ≤ 2 at study entry.
* Laboratory Requirements: (must be done within 7 days prior to first study drug dose)

Hematology: Absolute granulocytes (AGC) ≥ 1.0 x 109/L Platelets ≥ 50 x 109/L Chemistry: Serum creatinine ≤ 1.5 x UNL Bilirubin ≤ 1.5 x UNL AST (or ALT if AST ≤ 2.5 x UNL not available)

* Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL 10 - 14 days prior to therapy and repeated within 24 hours of starting study drug and must either commit to continued abstinence from heterosexual sexual intercourse or begin TWO acceptable methods of birth control, one highly effective methods and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide. In addition, sexually active WCBP must agree to ongoing pregnancy testing. Men must agree not to father a child and agrees to use a condom if his partner is of child bearing potential.
* Disease free of prior malignancies for ≥ 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast

Exclusion Criteria:

* Patients who fulfill any of the following criteria are not eligible for admission to the study:
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or lactating females. (Lactating females must agree not to breast feed while taking lenalidomide).
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Patients previously or currently receiving treatment with other anti-cancer therapy for CLL
* Lymphoproliferative disease other than CLL (includes patients with prolymphocytic leukemia, mantle cell lymphoma, and those who have transformed to a more aggressive lymphoma, or Richter's syndrome).
* Known hypersensitivity to thalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Any prior use of lenalidomide.
* Concurrent use of other anti-cancer agents or treatments.
* Known positive for HIV or infectious hepatitis, type A, B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine I Chen, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single site, Investigator initiated study. Patients gave informed consent according to institutional and university human experimentation committee requirements. Previously untreated B-cell CLL patients >/= 18 years of age were eligible if they met the eligibility criteria.
Pre-assignment Details: Study was halted and the protocol amended after severe toxicities were noted in the first 2 study patients when they were dosed as per the initial protocol dosing guidelines. Their data was not included in the analysis and additional 25 eligible patients were enrolled and their data was analyzed.
Groups:
- Lenalidiomide: Lenalidomide target dose of 10 mg PO OD X 3 weeks (days 1-21) followed by 1 week off therapy (days 22-28) on a 28-day cycle.
  Lenalidomide: Subjects will receive lenalidomide, starting at 2.5 mg daily x 3 weeks (days 1-21) and escalating up to a target dose of 10 mg daily X 3 weeks (days 1-21) followed by 1 week off therapy (days 22-28) on a 28 day cycle. Patients will be treated with lenalidomide until disease progression or 2 cycles past CR. (no maximum of cycles).
  Dose escalation beyond 10 mg daily to a maximum of 25 mgs daily was permitted for nonresponders.
Period: Overall Study
Arm/Group | Lenalidiomide
Started | 27 (The start date of the study was 25 August 2006.)
Completed | 25
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Groups:
- Lenalidiomide: Lenalidomide target dose of 10 mg PO OD X 3 weeks (days 1-21) followed by 1 week off therapy (days 22-28) on a 28-day cycle.
  Lenalidomide: Subjects will receive lenalidomide, starting at 2.5 mg daily x 3 weeks (days 1-21) and escalating up to a target dose of 10 mg daily X 3 weeks (days 1-21) followed by 1 week off therapy (days 22-28) on a 28 day cycle. Patients will be treated with lenalidomide until disease progression or 2 cycles past CR. (no maximum of cycles).
Arm/Group | Lenalidiomide
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] | 60 [33 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 16
Region of Enrollment [Number; unit: participants]
  Canada | 25

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Efficacy (Response Rate) of Oral Lenalidomide in the Treatment of Patients With Symptomatic, Previously Untreated, Chronic Lymphocytic Leukemia (CLL)
Description: The primary endpoint was objective response to lenalidomide (Complete response +Partial response) evaluated as per the revised 1996 National Cancer Institute Working Group Guidelines.
  Complete response: absence of lymphadenopathy and organomegaly by physical exam and radiology, absence of constitutional symptoms, normal CBC. Bone marrow to be done 2 months after the above criteria are met, must be normocellular, with <30% lymphocytes.
  Partial Response: ≥ 50% decrease in the peripheral blood lymphocytes from pre-treatment value, ≥ 50% reduction in lymphadenopathy and organomegaly by physical exam or on CT scan. one or more of the following: neutrophils ≥ 1.5 x109/L, platelets > 100 x109/L or 50% improvement over baseline, hemoglobin > 110 g/L or 50% improvement over baseline (without transfusion).
Time Frame: Patients will be treated with lenalidomide until disease progression or 2 cycles past CR (no maximum of cycles). Participants were followed upto 53.2 months for the final data analysis.
Population: Severe toxicities were seen in the first two patients enrolled on the initial protocol. The study was halted and the protocol amended to use a starting dose of lenalidomide 2.5 mg with monthly escalations to a target dose of 10 mg, extended tumor lysis prophylaxis and monitoring. 25 response evaluable patients were enrolled on the amended protocol.
Measure: Number; unit: participants
Arm/Group | Lenalidiomide
Number analyzed (Participants) | 25
participants
  Complete response | 5
  Partial response | 13
  Stable Disease | 6

2. Secondary Outcome: Percentage of Participants With Progression-free Survival (PFS) and Overall Survival (OS).
Description: Assess the time to disease progression and overall survival. (Progressive disease is defined as at least one of the following: more than or equal to 50% increase in the sum of the products of the greatest diameters of at least 2 lymph nodes on 2 consecutive determinations 2 weeks apart (at least one node must be ≥ 2 cm) or new palpable lymph nodes, more than or equal to 50% increase in the size of the liver and/or spleen as determined by measurement below the costal margin or appearance of palpable hepatomegaly or splenomegaly not previously present, more than or equal to 50% increase in the absolute number of circulating lymphocytes to at least 5.0 x109/L, OR transformation to a more aggressive histology (e.g. Richter's syndrome or prolymphocytic leukemia with >55% prolymphocytes)).
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidiomide
Number analyzed (Participants) | 25
percentage of participants
  Overall survival | 85.3 [71.1 to 100]
  Progression free survival | 64.6 [47.5 to 87.8]

ADVERSE EVENTS:
Description: CTCAE Version 3.0 was used for adverse event grading and categorizing
Arm/Group | Lenalidiomide
Serious Adverse Events (participants affected / at risk) | 17/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidiomide (N=25)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Disseminated Zoster (Infections and infestations) | 1 (1)
Coronary Artery disease (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Fever (General disorders) | 1 (1)
In-situ Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Thrombocytopenia (Investigations) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Community Acquired pneumonia (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Cytopenias (Investigations) | 1 (1)
Relapse of lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidiomide (N=25)
Tumor Flare (Blood and lymphatic system disorders) | 22 — Drug related
Fatigue (General disorders) | 18 — Drug related
Rash (Skin and subcutaneous tissue disorders) | 15 — Drug related
Myalgia (Musculoskeletal and connective tissue disorders) | 10 — Drug related
Pruritus (Skin and subcutaneous tissue disorders) | 8 — Drug related
Diarrhea (Gastrointestinal disorders) | 8 — Drug related
Constipation (Gastrointestinal disorders) | 6 — Drug related
Sensory neuropathy (Nervous system disorders) | 4 — Drug related
Leg edema (Blood and lymphatic system disorders) | 3 — Drug related
Dizziness (Nervous system disorders) | 3 — Drug related
Generalized Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 — Drug related
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 — Drug related
Elevated Creatinine (Investigations) | 11 — Drug related
Hypocalcemia (Investigations) | 11 — Drug related
Hypokalemia (Investigations) | 10 — Drug related
Hypophosphatemia (Investigations) | 10 — Drug related
Elevated AST or ALT (Investigations) | 9 — Drug related
Hypernatremia (Investigations) | 5 — Drug related
Hyponatremia (Investigations) | 4 — Drug related
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 — Drug related
Skin infection (Infections and infestations) | 4 — Drug related
Neutropenia (Investigations) | 18 — Drug related
Anemia (Blood and lymphatic system disorders) | 6 — Drug related
Thrombocytopenia (Investigations) | 7 — Drug related
Upper Respiratory/Sinus infection (Infections and infestations) | 2 — Drug related

LIMITATIONS AND CAVEATS:
Original study protocol used a starting lenalidomide dose of 10mg OD for 21days of a 28-day cycle, escalating weekly by 5mg to a target of 25mg daily. Toxicities reported with the first two enrolled patients lead to the current protocol amendment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less